CLINICAL TRIAL: NCT02878369
Title: Evaluation of Doppler Flow From the Femoral Artery as a Reflection of Cardiac Flow in a Vascular Fluid Test
Acronym: RER D
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC13_0486
Record Dates: First submitted 2016-08-22; First posted 2016-08-25 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Acute Circulatory Failure
Keywords: fluid replacement
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Doppler measurement of blood flow in the outflow tract of the left ventricle and the femoral artery,Reading blood pressures displayed on the monitor.

SUMMARY:
In order to identify the responding patients with vascular filling test, this research aims to compare the performance of the increased flow in the femoral artery to the performance of the blood pressure increase.

The reference measurement will increase cardiac output measured by ultrasound.

DETAILED DESCRIPTION:
It is notable that in the intensive care patient, the ultrasound measurement of cardiac flow is not always possible, especially in case of mechanical ventilation, often responsible for air interposed between the ultrasound probe and the heart, thus stopping the ultrasound. Use the blood pressure increase as a reflection of the increase in cardiac flow induced by fluid replacement is not a fully satisfactory alternative since its performance is at best just acceptable.

Flow measurement in the femoral artery could be an attractive alternative to the cardiac output measurement as:

* It is easy: the femoral vascular ultrasound is booming with resuscitators, including the laying of intravascular catheter or thrombosis diagnosis.
* It is painless: it is based on the application of the ultrasound probe on the root of the thigh for less than 5 minutes.
* It is not subject to limitations echogenicity by interposition of air (except in exceptional circumstances)
* It measures the same physiological parameter (arterial flow) as measuring ultrasound cardiac output (based on measurement of the flow at the outflow tract of the left ventricle).

Pathophysiology study, multicenter (conducted in three French ICUs), open, prospective in order to evaluate the flow doppler from the femoral artery as a reflection of cardiac flow in a vascular fluid test in patient with signs of acute circulatory failure in intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

Patient hospitalized in intensive care and affiliated to a social security system

* Intra-arterial catheter already in place and operational
* Stability blood pressure for 5 min (no change in mean arterial pressure> 10%, no increase in dose catecholamine)
* Presence of at least one sign of acute circulatory failure from:

  * Low blood pressure (mean arterial pressure <65 mmHg and / or systolic <90 mmHg)
  * tachycardia> 120 bpm without other obvious cause a circulatory failure
  * Oliguria <1 ml / kg during the last hour suggestive of circulatory failure
  * blood Hyperlactataemia> 2 mmol / l without other obvious cause a systemic circulatory failure (lactate will not be measured for the purposes of the study)
  * Smear
  * ongoing catecholamine Administration
  * Another sign justifying, according to the doctor in charge, vascular filling test (capillary refill time elongated, others ...)
* The doctor in charge has prescribed a fluid loading test, regardless of the needs of the study.

Non inclusion criteria:

Clear contraindication to the femoral artery Doppler (wound or burn the groin, for example)

* Complete occlusion of the femoral artery or 2 of the aorta requiring or having required a vascular bypass
* Pregnant woman
* Minor
* Major Trust

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: One hundred and twenty adult patients hospitalized in one of the participating ICUs, will be included (see the justification required number of subjects in "statistics") if
  * They are already carrying an intra-arterial catheter (femoral or radial).
  * They exhibit acute circulatory failure signs (see below)
  * The doctor in charge prescribed a vascular fluid replacement, regardless of the purposes of the study:
    * vascular fluid replacement
    * initiation or catecholamine
    * or increase (> 10%) of catecholamine dosage.
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
In the intensive care patient of acute circulatory failure signs, assess the increase of the femoral arterial flow (specifically its full-time speed, ΔRVAFitv measured by Doppler ultrasound) to identify responders this fluid replacement. | First patient enrollment: april 2014 - Study duration: 24 month - Patient follow-up: 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nantes, Nantes, France